CLINICAL TRIAL: NCT02544802
Title: Treatment of Primary Osteoarthritis of the Knee Joint With Autologous Mesenchymal Stem Cells
Brief Title: Mesenchymal Stem Cell Treatment for Primary Osteoarthritis Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Steminent Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB-VGH-201102
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ADMSCs (Experimental): Three intra-articular injections of ADMSCs at the dose of 8~10x10^6 cells/injection
  Interventions: Drug: Adipose-Derived Mesenchymal Stem Cells

INTERVENTIONS:
Drug: Adipose-Derived Mesenchymal Stem Cells

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of autologous adipose-derived mesenchymal stem cells (ADMSCs) treatment for patients with primary osteoarthritis knee. Three intra-articular injections of autologous ADMSCs will be performed to subjects at a weekly interval.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has bilateral Kellgren and Lawrence grade II-III primary osteoarthritis as determined by X-ray.
2. Subject's pain score is 8-13 points (Lequesne's index).
3. Ages between 50-70 years.
4. Signed informed consent from the subject.
5. Female subjects should be post-menopausal women

Exclusion Criteria:

1. Subject infected with hepatitis B, hepatitis C, HIV, syphilis or HTLV.
2. Subject not suitable for liposuction surgery.
3. Subject with hypersensitivity/allergy to anesthetic.
4. Subject's creatinine values higher than 1.6mg/dl.
5. Subject with body mass index, BMI over 30.
6. Subject's studied knee treated with intra-articular injection therapy within 6 months prior to screen.
7. Subject has undergone surgery on either side of knee, including fracture surgery, arthroscopic surgery, meniscus repair surgery, or cruciate ligament reconstruction surgery.
8. Subject enrolled in any other cell therapy studies within the past 30 days.
9. Subject who the investigator considers inappropriate for the clinical trial due to any other reasons than those listed above.
10. Subject has a history of gouty arthritis, septic arthritis, rheumatoid arthritis and any other autoimmune arthritis of the knee joint.
11. Subject has had major medical problems in vital organs, such as; heart, liver, kidney, or lung.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-06; Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Safety of intra-articular injection of autologous ADMSCs by incidence of adverse events and alterations in vital signs, blood chemistry profiles, complete blood count, urinalysis, and also the physical examination of the knees. | 12 months

SECONDARY OUTCOMES:
Clinical assessment of visual analogue scale (VAS) | 12 months
Clinical assessment of Short Form 36 questionnaire (SF-36) | 12 months
Clinical assessment of Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 12 months
Clinical assessment of Hospital for Special Surgery (HSS) Knee Score | 12 months
Clinical imaging assessment of knee X-ray | 12 months
Clinical imaging assessment of MRI of the knee | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan